CLINICAL TRIAL: NCT05558839
Title: The Effect of Exercise and Cognitive Training on the Physical Fitness, Fall, and Cognition Among Community-dwelling Older Adults With Dementia.
Brief Title: The Effect of Exercise and Cognitive Training on Community-dwelling Older Adults With Dementia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-02-022B
Record Dates: First submitted 2022-09-07; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Dementia; Exercise; Fall; Cognitive Training
MeSH Terms: conditions — Dementia; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study adopted a quasi-experimental study design involving single-group pretest-posttest. The research participants were 41 community-dwelling older adults with mild or moderate dementia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise training (Experimental): Physiotherapists prescribed and delivered interventions in the exercise arm. Each exercise session began with a 5-minute warm up and stretching, followed by 15-minute Aerobic exercises, 15-minute of resistance training, 10-minute of agility and balance training, and 5-minute of cooling down.
  Interventions: Behavioral: A 12-week weekly sports and cognitive training intervention.
- cognitive training (Experimental): Board game teachers who have more than 5 years of community teaching experience prescribed and delivered interventions in the cognitive arm.
  Each cognitive session uses different board games to strengthen training for different cognitive aspects.
  Interventions: Behavioral: A 12-week weekly sports and cognitive training intervention.

INTERVENTIONS:
Behavioral: A 12-week weekly sports and cognitive training intervention. — A 12-week weekly sports and cognitive training intervention was provided to the participants. The training, 2 hours each week, involved 1 hour of sports training and 1 hour of cognitive training.

SUMMARY:
This study aimed to explore the effects of an exercise and cognitive training intervention on the physical fitness, fall, and cognitive functions of community-dwelling older adults with dementia. The exercise and cognitive training intervention of this study promoted physical fitness, reduced chance of falling, and improved the cognitive functions of community-dwelling older adults with dementia. In addition, the score of risk of falling reduced.

DETAILED DESCRIPTION:
Taiwan has become an aged society, and its population with dementia increases rapidly. Older adults with dementia have unfavorable balance ability and may lack muscle strength; consequently, their probability of falling is twice as high as that of healthy older adults, and their probability of falling and being hospitalized is three times that for general healthy older adults. Compared to European countries and the United States, Taiwan has limited studies on older adults with dementia regarding effects of exercise and cognitive intervention. To develop an intervention for older adults with dementia that integrates exercise and cognitive training to promote or maintain their physical fitness and cognitive function to reduce their risk of falling is critical.

This study adopted a quasi-experimental study design involving single-group pretest-posttest. The research participants were 41 community older adults with mild or moderate dementia. Participants were recruited from 5 community-based dementia care centers in Taipei City. A 12-week weekly sports and cognitive training intervention was provided to the participants. The training, 2 hours each week, involved one hour of sports training and one hour of cognitive training.

Physiotherapists prescribed and delivered interventions in the exercise arm. Each exercise session began with a 5-minute warm up and stretching, followed by 15-minute Aerobic exercises, 15-minute of resistance training, 10-minute of agility and balance training, and 5-minute of cooling down.

Board game teachers who have more than 5 years of community teaching experience prescribed and delivered interventions in the cognitive arm.

Each cognitive session uses different board games to strengthen training for different cognitive aspects.

Before and after the intervention, data of the participants' functional physical fitness, their scores of the STRATIFY Falls Risk Assessment, and their scores of the Montreal Cognitive Assessment were collected as the outcome indicators. A paired t test was used to analyze the results of the intervention. This study aimed to explore the effects of an exercise and cognitive training intervention on the physical fitness, fall, and cognitive functions of community older adults with dementia.

ELIGIBILITY:
Inclusion Criteria:

* The list of dementia cases under the supervision of the Taipei City Government Health Bureau, who are over 65 years of age and have been diagnosed with mild to moderate dementia.
* Those who can participate in sports activities.
* Those who can communicate in both Chinese and Taiwanese, have self-determination ability and can clearly express their wishes.

Exclusion Criteria:

* Those who have exercise contraindications due to medical reasons.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
functional physical fitness | 14 weeks (Before and after interventions)
  Physiological measurements:
  * The 30 second chair stand test is for testing leg strength and endurance in older adults. This requires people to repeatedly stand up from and sit down on a chair for 30 seconds. The number of stands is recorded. This reﬂects lower body strength.
  * The handgrip strength test is to measure the maximum isometric strength of the hand and forearm muscles.
  * The 8-foot up-and-go test is used to measure balance, agility, and speed while walking or moving.
Falls risk assessment | 14 weeks (Before and after interventions)
  We reported fall risk was assessed with the STRATIFY assessment tool(St. Thomas Risk Assessment Tool in Falling Elderly Inpatients) by questionnaire.
  Falls risk assessment tool is used to identify fall risk factors for falls in the elderly and to predict the chance of falling.
  This tool comprises five items addressing risk factors: past history of falling, patient agitation, visual impairment, incontinence, transfer and mobility. The STRATIFY score range from 0 to 5 points and the predictive cut off of risk of falling is a score ≥ 2 points.
Cognitive Assessment | 14 weeks (Before and after interventions)
  We reported cognitive assessment was assessed with the Taiwan version of Montreal Cognitive Assessment (MoCA-T) by questionnaire.
  The Montreal Cognitive Assessment (MoCA) is a test used by healthcare providers to evaluate people with memory loss or other symptoms of cognitive decline. The MoCA contains 30 questions and takes around 10 to 12 minutes to complete. The MoCA checks different types of cognitive or thinking abilities. These include: orientation, short-term memory/delayed recall, executive function/visuospatial ability, language, abstraction, animal naming, attention, and clock-drawing test. The MoCA test uses a 30-point scale and take only 10 to 12 minutes. to complete. Scores on the MoCA range from zero to 30. A score of 26 and higher is considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Hui-Wen, M.D., Principal Investigator — member
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan